CLINICAL TRIAL: NCT06772337
Title: the Risk Prediction Model of Major Adverse Cardiovascular Events After PCI in Patients With Acute Myocardial Infarction Based on Multimodal Machine Learning and the Effect of Digital Therapeutics for Cardiac Rehabilitation
Brief Title: Effect of Digital Therapeutics for Cardiac Rehabilitation in Patients With Acute Myocardial Infarction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chen Leilei, Director, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTCR
Record Dates: First submitted 2024-12-31; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Acute Myocardial Infarction; Cardiac Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digitalized Cardiac Rehabilitation Group (Experimental Group) (Experimental): Intervention group patients received in-hospital cardiac rehabilitation during their hospital stay and a digital cardiac rehabilitation program after discharge.
  Interventions: Behavioral: digital cardiac rehabilitation
- Regular Treatment Group (Control Group) (Experimental): The patients in the control group received in-hospital cardiac rehabilitation during their hospitalization, and after discharge, they conducted cardiac rehabilitation training at home by themselves and returned to the hospital for regular follow-up.
  Interventions: Behavioral: Regular Treatment

INTERVENTIONS:
Behavioral: digital cardiac rehabilitation — Intra-hospital cardiac rehabilitation: For patients after PCI, reasonable dietary intervention, conventional drug treatment and conventional rehabilitation are given, without lower extremity power bike and respiratory training.Outside-hospital cardiac rehabilitation: The experimental group received conventional treatment and secondary prevention drugs recommended by the current guidelines, and carried out supervised digital cardiac rehabilitation on this basis.Doctors prescribe progressive aerobic exercise (walking) through mobile phone apps or computer terminals. Patients will train with wearable devices that can monitor physiological parameters in real time through the mobile phone FREE Rehabilitation APP.
  Arms: Digitalized Cardiac Rehabilitation Group (Experimental Group)
Behavioral: Regular Treatment — Intra-hospital cardiac rehabilitation: For patients after PCI, reasonable dietary intervention, conventional drug treatment and conventional rehabilitation are given, without lower extremity power bike and respiratory training.Out-of-hospital cardiac rehabilitation: Receiving conventional treatment and secondary prevention drugs recommended by current guidelines, nutritional diet and lifestyle guidance, and establishing a WeChat group as a postoperative follow-up contact method.Outside-hospital cardiac rehabilitation: The experimental group received conventional treatment and secondary prevention drugs recommended by the current guidelines, and carried out supervised digital cardiac rehabilitation on this basis.Doctors prescribe progressive aerobic exercise (walking) through mobile phone apps or computer terminals. Patients will train with wearable devices that can monitor physiological parameters in real time through the mobile phone FREE Rehabilitation APP.
  Arms: Regular Treatment Group (Control Group)

SUMMARY:
This study adopts a multicenter, open-label, randomized controlled clinical study, with Jiangsu Provincial People's Hospital as the leading unit, and the other 13 hospitals as cooperative units.

DETAILED DESCRIPTION:
It uniformly deploys an integrated cardiac rehabilitation management platform from the hospital to outside the hospital. Based on this platform, precise cardiac rehabilitation for myocardial infarction patients based on continuous dynamic physiological data is carried out. A total of 160 myocardial infarction patients after PCI who will undergo digital therapy cardiac rehabilitation are randomly divided into a digital cardiac rehabilitation group (experimental group) and a conventional treatment group (control group) at a ratio of 1:1 using a computer random sequence method, with 80 patients included in each group.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets the diagnostic criteria for AMI in the "Diagnosis and Treatment Guidelines for Acute ST-Segment Elevation Myocardial Infarction (2019)" and undergoes PCI for the first time;
* The age is between 18 and 75 years old;
* The left ventricular ejection fraction (LVEF) is 35% - 50%;
* The patient has normal cognition and can cooperate with the test;
* The patient signs the informed consent and the agreement to participate in this study.

Exclusion Criteria:

* Symptom-limited cardiopulmonary exercise test (treadmill) contraindications:

  1. Uncontrolled acute coronary syndrome;
  2. Acute heart failure;
  3. Symptomatic severe aortic stenosis, severe aortic coarctation or descending aortic aneurysm;
  4. Acute aortic dissection;
  5. Acute myocarditis, pericarditis or endocarditis;
  6. Symptomatic or hemodynamically unstable severe arrhythmia;
  7. Severe bradyarrhythmia;
  8. Acute pulmonary embolism and pulmonary infarction;
  9. Acute respiratory failure;
  10. Uncontrolled asthma;
  11. Peripheral oxygen saturation < 88% at rest or heart rate > 120 beats/min;

  s. Uncontrolled hypertension: systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg; t. Recent stroke or transient ischemic attack; u. Intermuscular venous thrombosis of the lower extremities; v. Orthopedic injury that hinders walking; w. Mental abnormality; x. Those who cannot cooperate;
* Patients who have not completed revascularization treatment or have planned revascularization within one year;
* Pregnant or lactating patients, or those who plan to become pregnant within one year;
* Patients who have received mechanical circulatory support treatment (such as intra-aortic balloon counterpulsation, Impella, ECMO, etc.) or tracheal intubation;
* Patients with a history of non-ischemic cardiomyopathy such as viral myocarditis or dilated cardiomyopathy, hypertrophic cardiomyopathy, peripartum cardiomyopathy, etc.;
* Patients with moderate or severe valvular heart disease or a history of valve replacement;
* Severe liver function abnormality (ALT ≥ 3 times the upper limit of the normal range) or renal function abnormality (eGFR < 60 mL/min/1.73 m2);
* Patients with diseases such as malignant tumors and an expected lifespan of less than one year;
* Those who cannot use a smartphone for various reasons and are inconvenient to communicate with the management team;
* Those who are participating in other clinical trials;
* The researcher believes that there are any other clinical conditions that are not suitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | 12 months
  The test requirements refer to the guidelines formulated by the American Thoracic Society. Instruct the patient to walk back and forth on a 30-meter-long corridor at the fastest speed. Once there are obvious symptoms such as chest tightness, dizziness, and breathing difficulties, the experiment should be stopped immediately, and the walking distance of the patient within 6 minutes should be detected and recorded after the experiment.
maximal oxygen uptake(VO2 max) | 12 months
  maximal oxygen uptake(VO2 max) is measured by Cardiopulmonary exercise testing (CPET). CPET refers to a method of examination that, under a gradually increasing exercise load, measures a series of indicator changes in the human body, including gas metabolism, heart rate, blood pressure, blood oxygen saturation, and electrocardiogram, from the resting state to the maximum exertion state during exercise and then back to the resting state. It records the corresponding symptoms that occur in the subjects during the testing process, objectively reflecting the physiological and pathological changes and the degree of functional impairment that occur at different load levels, thereby comprehensively evaluating the overall function and reserve capacity of organ systems such as the heart and lungs. The protocol used in this study is a symptom-limited incremental exercise test using a treadmill.
electrocardiogram | 12 months
  Wear a wearable device, and the monitoring time is from 8:00 am to 8:00 am the next day. Collect physiological signals such as electrocardiogram to evaluate heart rate variability and activity levels.
breathing patterns | 12 months
  Wear a wearable device, and the monitoring time is from 8:00 am to 8:00 am the next day. Collect physiological signals such as breathing to evaluate breathing patterns, sleep breathing events, sleep stages.
blood oxygen | 12 months
  Wear a wearable device, and the monitoring time is from 8:00 am to 8:00 am the next day. Collect physiological signals such as blood oxygen to evaluate breathing patterns, sleep breathing events, sleep stages.
The left ventricular ejection fraction ( LVEF) | 12 months
  The patient's left ventricular ejection fraction ( LVEF) is detected by echocardiography. The patient is in the supine position, and the probe scans the parasternal long-axis view of the left ventricle, the apical four-chamber view, the two-chamber view, the short-axis view of the ventricle, etc. The left ventricular ejection fraction ( LVEF) is determined. The value are obtained by calculating the average of three consecutive cardiac cycles in the apical four-chamber view using the modified Simpson's rule.

SECONDARY OUTCOMES:
Barthel Index | 12 months
  Barthel Index: The ability of daily living self-care is evaluated by the Barthel Index, which consists of 10 items, including eating, bathing, grooming, dressing, bowel control, bladder control, toileting, transfer from bed to chair, walking, and going up and down stairs. The total score ranges from 0 to 100. The higher the score, the better the self-care ability. A score of 100 indicates complete self-care.
score of the Generalized Anxiety Disorder 7-item scale (GAD-7) | 12 months
  Anxiety is assessed using the Generalized Anxiety Disorder 7-item scale (GAD-7). A total score of ≥5 in the assessment result is positive, indicating the possible presence of anxiety. Among them, a score of 5 - 9 may indicate mild anxiety, 10 - 14 may indicate moderate anxiety, and 15 - 21 may indicate severe anxiety.
score of the Patient Health Questionnaire-9 (PHQ-9) | 12 months
  Depression is assessed using the Patient Health Questionnaire-9 (PHQ-9). A total score of ≥5 in the assessment result is positive, indicating the possible presence of depressive mood. Among them, a score of 5 - 9 may indicate mild depression, 10 - 14 may indicate moderate depression, and 15 - 27 may indicate severe depression.
incidence rate of Major Adverse Cardiovascular Events (MACE) | 12 months
  Major Adverse Cardiovascular Events include heart failure, cardiovascular death, arrhythmia, atrial fibrillation, ventricular tachycardia, all-cause mortality, readmission, cardiogenic shock, target vessel revascularization, new or worsening myocardial infarction, non-fatal stroke, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangqing Kong, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China